CLINICAL TRIAL: NCT06151925
Title: Laminaria Tents Versus Vaginal Prostaglandin in Cervical Ripening in Term Induction of Labor With Unfavorable Cervix:A Randomized Controlled Trial
Brief Title: Laminaria Tents Versus Vaginal Prostaglandin in Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU M D 63/2021
Record Dates: First submitted 2022-05-25; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2021-05

CONDITIONS: Labor Onset and Length Abnormalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Laminaria tents group (Active Comparator): Laminaria tent used to be inserted in cervix and left for 6-12 hours
  Interventions: Device: Laminaria; Drug: Vaginal prostaglandin
- vaginal prostaglandin group (Placebo Comparator): Misoprostol 25 mcg inserted for one or multiple doses
  Interventions: Device: Laminaria; Drug: Vaginal prostaglandin

INTERVENTIONS:
Device: Laminaria — mechanical method for induction of labor
Drug: Vaginal prostaglandin — Vaginal prostaglandin for ripening
  Other Names: Vagiprost

SUMMARY:
Mechanical methods used for induction of labor received a great attention nowadays due to the serious side effects of the pharmacological methods. Hygroscopic dilators are considered important subtype of these mechanical methods. One of them is Laminaria which is a synthetic type of sea algae that induces cervical dilation by absorbing water from the cervix and gradually increasing in thickness. The current study will compare the effectiveness and safety of laminiria and vaginal prostaglandins in induction of labor in women with unfavorable cervix.

DETAILED DESCRIPTION:
A new method for induction of labor to be studied

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with:

  * Age 18-45 years.
  * Live fetus with cephalic presentation.
  * Normal non-stress test with reassuring features (baseline heart rate 110-160 beats/min, baseline variability 5-25 beats/minute, and no decelerations) (National Institute for Health and Clinical Excellence 2017).
  * Gestational age of 37 weeks or more (Middleton et al. 2020).
  * Fetal weight less than 4 kilograms.
  * Bishop score less than 6 (Navve et al. 2017).
  * No labor pains.
  * No contraindications for vaginal delivery

Exclusion Criteria:

* o Presence of fetal distress.

  * Presence of thick meconium-stained amniotic fluid
  * Presence of fever, chorioamnionitis, or vaginal bleeding before intervention.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 90 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
o Bishop Score and cervical dilatation | 2 YEARS
  Tool to assess cervical status

SECONDARY OUTCOMES:
o Induction time to active phase of labor. | 2 YEARS
  Time between start and 5cm dilatation
o Induction time to delivery time. | 2 YEARS
  Time between start to delivery

OTHER OUTCOMES:
o Cesarean frequency rate | 2 YEARS
  Number of needed cs
o Intrapartum complications | 2 YEARS
  Any complicated case

CONTACTS AND LOCATIONS:
Overall Officials: Maya AbdelRazek, MD, Principal Investigator — Lecturer of obstetrics and gynecology - Ain Shams University
Locations (1):
- Ain Shams University Faculty Of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
It will be available once approved
Supporting Information: Study Protocol
Time Frame: Within one month from now
Access Criteria: Open access